CLINICAL TRIAL: NCT06827808
Title: The Effect of Team-Based Learning on Nursing Students' Skill Acquisition in Fundamental Nursing Education: a Randomized Controlled Trial
Brief Title: The Effect of Team-Based Learning on Nursing Students' Skill Acquisition in Fundamental Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Gamze Bolattürk, Doctor Research Assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Gamze Bolattürk
Record Dates: First submitted 2025-02-01; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Team Based Learning; Nursing Skills; Academic Success

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled single-blind quasi-experimental research design.
Who Masked: Participant
Masking Description: In the randomization process, those who meet the criteria for inclusion in the sample and accept to participate in the study do not know that they will be included in the intervention group or the control group, so it will be single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Team Based Learning (Experimental): The experimental group students were first administered iRAT. After iRAT, the students were divided into groups and formed teams and worked together for approximately 30 minutes to critique the same skill and then repeated it. Then, tRAT, which included the same questions as iRAT questions and lasted 10 minutes, was administered. In the tRAT application, students held group discussions to reach a consensus on the answers to the MCQs. When the students in the team found a suitable answer different from the answer they had chosen, they discussed the question again until they agreed on a new answer. After the tRAT was completed, the instructor discussed the correct answers to the questions with all groups and shared the group scores.
  Interventions: Other: Team based learning
- Control Group (No Intervention): Control group students individually practiced the relevant nursing skills on models in the laboratory during the lesson.

INTERVENTIONS:
Other: Team based learning — The intervention planned within the scope of the research is a team-based learning method. Students in the intervention group taking the nursing fundamentals course will be formed into small groups in the nursing skills laboratory. The groups will remain the same throughout the six modules. First, students will be asked to solve the iRAT multiple-choice question set prepared on the relevant module skill. Then, students will be provided with the skill repetition in the determined groups. Then, they will be asked to discuss until they reach a consensus as a group and solve the tRAT, which includes the same multiple-choice question set as the iRAT.
  Arms: Team Based Learning

SUMMARY:
Nursing education is a practical education where theoretical knowledge is combined with laboratory and clinical skills. Skill practices that students should gain during nursing education constitute one of the most important components of the nursing profession. New methods are gaining popularity due to the fact that traditional learning methods do not attract the attention of today's student profile and cannot meet the needs at the desired level. This situation has led to the emergence and spread of active teaching and learning methods, including the cooperative learning approach. Since the learner is directly involved in the learning process in cooperative learning, active participation contributes to the development of the student in many ways. Team-Based Learning (TBL), one of the cooperative teaching methods, is a teaching method that encourages students to think critically and solve clinical problems not only individually but also as a team, and also develops problem solving, effective teamwork and communication skills. TBL is an interactive teaching strategy designed to increase student engagement. Introduced in higher education in the late 1970s, this method is based on constructive learning theory, in which students develop new personal and mental frameworks based on their prior knowledge. TBL is a method that encourages the development of student competencies, including self-directed learning, critical thinking, analysis and application, as well as team collaboration and interpersonal skills. TBL is a teaching strategy planned to be implemented in multiple stages. TBL begins with students' pre-lesson preparation, students apply preparation assurance tests individually and as a team, and the method ends with the evaluation and application of course concepts by the instructor. It is thought that the use of the TBL method in nursing education will contribute to the development of important clinical skills by using clinical experience, knowledge, and problem-solving skills. In the literature, it has been reported that TBL is an effective teaching strategy in improving problem-solving ability, knowledge and clinical performance, that it promotes learning and contributes significantly to the academic performance of students. One of the important factors that should be evaluated regarding the clinical competence of nursing students is their academic success level. Academic success can be measured by different methods including problem-solving skills, clinical competence, general grade point average and skill assessment exams (OSCE). OSCE (Objective Structured Clinical Examination) is among the methods used to evaluate the academic success of nursing students. This study aimed to evaluate the effect of TBL on the academic success of students in skills training.

ELIGIBILITY:
Inclusion Criteria:

* first time learning nursing care skills
* volunteering to participate in the study

Exclusion Criteria:

* not attending class and being absent
* not wanting to participate in research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Individual Readiness Assurance Test (iRAT) | At the end of the 45 minute lesson
  Individual Readiness Assurance Test (iRAT) is the first step in which students are asked to solve a prepared list of Multiple Choice Questions (MCQ) individually. The experimental group students were first given iRAT, which lasted 10 minutes. After the iRAT application, the students were not given the answers to the questions.

SECONDARY OUTCOMES:
Team Readiness Assurance Test (tRAT) | 45 minutes after iRAT
  After the Individual Readiness Assurance Test (iRAT), students are distributed into small teams and solve the same set of MCQs again through group discussion until a consensus is reached, representing the Team Readiness Assurance Test (tRAT). After the iRAT, students took a 15-minute break. After the break, students were divided into teams and worked together for about 30 minutes to critique and revise the same skill. Then, tRAT, which included the same questions as the iRAT questions and lasted for 10 minutes, was administered. In the tRAT application, students conducted group discussions to reach a consensus on the answers to the MCQs. When students in the team found a suitable answer different from the answer they had chosen, they discussed the question again until they agreed on a new answer. After the tRAT was completed, the instructor discussed the correct answers to the questions with all the groups and shared the group scores.
OSCE (Objective Structured Clinical Examination) | 8 weeks after starting the study
  OSCE is a station-based, reliable and impartial assessment tool in which students demonstrate specific skills in a simulated environment over a period of time. In the study, checklists of drug administration, injection administration, hygiene administration, respiratory administration, movement administration and nutrition administration skills in six modules were used to assess the skill levels of students. The lowest score that can be obtained from the skill checklists is "0" and the highest score is "100".

CONTACTS AND LOCATIONS:
Overall Officials: Doctor Research Assistant, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No